CLINICAL TRIAL: NCT00344578
Title: Clinical Outcomes After AcrySof® ReStor IOL Surgery in Faculty Practice at UTSW Medical Center at Dallas: A Retrospective Review
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Adam Fedyk, MD, UTSW Medical Center at Dallas
Other Study IDs: Fedyk001
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2006-06

CONDITIONS: Outcomes Following Restor IOL Lens Implant
Keywords: Higher Order Abberations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Restor IOL

SUMMARY:
To evaluate the clinical outcomes of AcrySof® ReSTOR® IOL for the Faculty Practice at UTSW Medical Center at Dallas

DETAILED DESCRIPTION:
The AcrySof® ReSTOR® intraocular lens (IOL) is the latest advance in vision surgery. This IOL has been uniquely designed to improve vision throughout the entire visual spectrum, up close, far away and everything in-between. Thus, giving cataract patients their best chance ever to function free of glasses.

The pre-operative and post-operative data from ReSTOR® IOL implant cataract surgeries will be analyzed to determine whether the desired outcome was achieved, i.e. excellent vision with no correction. Variables to be studied include patient age, gender, number of ReSTOR® IOL implants, ocular comorbidities, preoperative and postoperative corrected and uncorrected visual acuities, keratometry readings, and corneal topography readings. A patient survey will also be sent to patients having undergone the surgery to measure their level of satisfaction.

Project Goals: The ultimate outcome of this project is to learn more insight on the following:

1. Visual acuity with and without correction of distance and near at 3-6 months
2. Percent of patients requiring keratorefractive surgery
3. Ocular comorbidity subgroup analysis
4. Monocular implantation subanalysis (prior to LASIK)
5. Comparison of post-op spherical equivalent to target refraction
6. Posterior capsule opacity that may be treated with laser procedure known as a YAG laser capsulotomy?
7. Subjective patient satisfaction
8. Validated questionnaire assessing visual function and quality of life

ELIGIBILITY:
Inclusion Criteria:

All patients of any race and sex between the ages of 18-90 years of age who have undergone ReSTOR® IOL cataract surgery will be recruited in this retrospective project.

Exclusion Criteria:

Patients who underwent conventional IOL cataract extraction surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients of any race and sex between the ages of 18-90 years of age who have undergone ReSTOR® IOL cataract surgery will be recruited in this retrospective project.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2006-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
1)Visual acuity with and without correction of distance and near at 3-6 months

SECONDARY OUTCOMES:
Percent of patients requiring keratorefractive surgery
Ocular comorbidity subgroup analysis
Monocular implantation subanalysis (prior to LASIK)
Comparison of post-op spherical equivalent to target refraction
Posterior capsule opacity that may be treated with laser procedure known as a YAG laser capsulotomy?
Subjective patient satisfaction
Validated questionnaire assessing visual function and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Adam Fedyk, MD, Principal Investigator — UTSW Medical Center at Dallas; Vinod Mootha, MD, Study Director — UTSW Medical Center at Dallas; James McCulley, MD, Study Chair — UTSW Medical Center at Dallas
Locations (2):
- United States (2):
  - Aston Ambulatory Care Center, Dallas, Texas
  - UTSW Medical Center at Dallas, Dallas, Texas